CLINICAL TRIAL: NCT05239312
Title: Antibiogram and Biofilm Formation of Bacteria Causing Prosthetic Joint Infections Isolated From Assiut University Hospital
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amina Abd El Aal Mohammed Abd El Aal Makhlouf, Assistant lecturer, Assiut University
Other Study IDs: Antibiogram and biofilm in PJI
Record Dates: First submitted 2021-11-14; First posted 2022-02-14 (Actual); Last update posted 2022-02-14 (Actual); Status verified 2022-02

CONDITIONS: Prosthetic Joint Infection
MeSH Terms: interventions — Anti-Infective Agents

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with prosthetic joint infection
  Interventions: Drug: Antimicrobial

INTERVENTIONS:
Drug: Antimicrobial — Implementation of antimicrobial protocol for empirical treatment which will be done according to the results of antibiotic susceptibility
  Other Names: Implementation of infection prevention and control policies

SUMMARY:
1. Setting of antibiogram in orthopedic department
2. Evaluate the production of biofilm in bacteria isolated from specimens phenotypically and genotypically.

DETAILED DESCRIPTION:
Increased use of total joint arthroplasties will naturally result in a related increase in the number of prosthetic joint infections (PJIs).

PJI is a disastrous complication of orthopedic surgery, frequently leading to prolonged morbidity and increased mortality. Moreover, therapy for PJI is associated with enormous costs.

PJI results from numerous factors that lead to inability of periprosthetic immune cells to protect implant surfaces and tissues from bacterial colonization.

The most destabilizing factor is the ability of bacteria to adhere to and survive on virtually all natural and synthetic surfaces.

Once firmly attached to the surface of an implant, the microorganisms initiate "biofilm" formation, which is a complex of microbial cells embedded in an extracellular matrix composed of proteins, extracellular DNA, and exopolysaccharides, providing protection for bacteria and making them extremely resistant to the immune system and antibiotic.

An ineffective empiric antibiotic regimen can be harmful to patients while unnecessary broad-spectrum antibiotics lead to increased resistance. However, healthcare providers often select an antibiotic regimen before bacterial antibiotic sensitivities are available.

The Clinical and Laboratory of Standards Institute publishes the M39 Analysis and Presentation of Cumulative Antimicrobial Susceptibility Test Data; Approved Guideline, which is a referenced guideline on how to create antibiograms.

The antibiogram has multiple uses, including providing guidance for empiric antibiotic therapy, monitoring changes in resistance over time, assisting in formulary decisions and supports antimicrobial stewardship programs to reduce multidrug resistant organisms and the risks of adverse drug events.

ELIGIBILITY:
1. Inclusion criteria:

   * Age above 18 years old
   * no intraarticular surgery of the respective joint prior to the index surgery.
2. Exclusion criteria:

   * Age below 18 years old
   * If the patient had any intraarticular surgery prior to the primary arthroplasty in the respective joint.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will be conducted on 90 informed individuals (according to guidelines of ethical committee of faculty of medicine , Assuit University )
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2022-03 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Antibiogram for PJI | 18 months
  Percentages of different bacterial species causing prosthetic joint infection and their Antimicrobial sensitivity pattern.

SECONDARY OUTCOMES:
Biofilm formation | 18 months
  Percentage of different bacteria responsible for biofilm formation

REFERENCES:
- [Background] Gallo J, Nieslanikova E. Prevention of Prosthetic Joint Infection: From Traditional Approaches towards Quality Improvement and Data Mining. J Clin Med. 2020 Jul 11;9(7):2190. doi: 10.3390/jcm9072190. PMID 32664491
- [Background] Fischbacher A, Borens O. Prosthetic-joint Infections: Mortality Over The Last 10 Years. J Bone Jt Infect. 2019 Sep 17;4(4):198-202. doi: 10.7150/jbji.35428. eCollection 2019. PMID 31555507
- [Background] Natsuhara KM, Shelton TJ, Meehan JP, Lum ZC. Mortality During Total Hip Periprosthetic Joint Infection. J Arthroplasty. 2019 Jul;34(7S):S337-S342. doi: 10.1016/j.arth.2018.12.024. Epub 2018 Dec 24. PMID 30642705
- [Background] Musil D, Snorek M, Gallo J, Jahoda D, Stehlik J. [Economic Analysis of the Costs of Hospital Stay of Patients with Infection as a Complication of Total Replacements - Part 2: Total Hip Arthroplasty]. Acta Chir Orthop Traumatol Cech. 2019;86(4):241-248. Czech. PMID 31524584
- [Background] Musil D, Snorek M, Gallo J, Jahoda D, Stehlik J. [Economic Analysis of the Costs of Hospital Stay of Patients with Infection as a Complication of Total Replacements - Part 1: Total Knee Arthroplasty]. Acta Chir Orthop Traumatol Cech. 2019;86(3):173-180. Czech. PMID 31333180
- [Background] Puhto T, Puhto AP, Vielma M, Syrjala H. Infection triples the cost of a primary joint arthroplasty. Infect Dis (Lond). 2019 May;51(5):348-355. doi: 10.1080/23744235.2019.1572219. Epub 2019 Apr 2. PMID 30938200
- [Background] Davidson DJ, Spratt D, Liddle AD. Implant materials and prosthetic joint infection: the battle with the biofilm. EFORT Open Rev. 2019 Nov 5;4(11):633-639. doi: 10.1302/2058-5241.4.180095. eCollection 2019 Nov. PMID 31754470
- [Background] Arciola CR, Campoccia D, Montanaro L. Implant infections: adhesion, biofilm formation and immune evasion. Nat Rev Microbiol. 2018 Jul;16(7):397-409. doi: 10.1038/s41579-018-0019-y. PMID 29720707
- [Background] Baker P, Hill PJ, Snarr BD, Alnabelseya N, Pestrak MJ, Lee MJ, Jennings LK, Tam J, Melnyk RA, Parsek MR, Sheppard DC, Wozniak DJ, Howell PL. Exopolysaccharide biosynthetic glycoside hydrolases can be utilized to disrupt and prevent Pseudomonas aeruginosa biofilms. Sci Adv. 2016 May 20;2(5):e1501632. doi: 10.1126/sciadv.1501632. eCollection 2016 May. PMID 27386527
- [Background] Orazi G, O'Toole GA. "It Takes a Village": Mechanisms Underlying Antimicrobial Recalcitrance of Polymicrobial Biofilms. J Bacteriol. 2019 Dec 6;202(1):e00530-19. doi: 10.1128/JB.00530-19. Print 2019 Dec 6. PMID 31548277
- [Background] Paul M, Shani V, Muchtar E, Kariv G, Robenshtok E, Leibovici L. Systematic review and meta-analysis of the efficacy of appropriate empiric antibiotic therapy for sepsis. Antimicrob Agents Chemother. 2010 Nov;54(11):4851-63. doi: 10.1128/AAC.00627-10. Epub 2010 Aug 23. PMID 20733044
- [Background] Kuti EL, Patel AA, Coleman CI. Impact of inappropriate antibiotic therapy on mortality in patients with ventilator-associated pneumonia and blood stream infection: a meta-analysis. J Crit Care. 2008 Mar;23(1):91-100. doi: 10.1016/j.jcrc.2007.08.007. PMID 18359426
- [Background] Klinker KP, Hidayat LK, DeRyke CA, DePestel DD, Motyl M, Bauer KA. Antimicrobial stewardship and antibiograms: importance of moving beyond traditional antibiograms. Ther Adv Infect Dis. 2021 May 5;8:20499361211011373. doi: 10.1177/20499361211011373. eCollection 2021 Jan-Dec. PMID 33996074
- [Background] Mitchell SL, Shaffer ML, Loeb MB, Givens JL, Habtemariam D, Kiely DK, D'Agata E. Infection management and multidrug-resistant organisms in nursing home residents with advanced dementia. JAMA Intern Med. 2014 Oct;174(10):1660-7. doi: 10.1001/jamainternmed.2014.3918. PMID 25133863